CLINICAL TRIAL: NCT05032170
Title: In Vivo Accuracy of Two Intraoral Scanning Systems in Detecting Two Inter-foraminal Implants in the Edentulous Mandible.
Brief Title: Intraoral Scanning Accuracy in the Edentulous Mandible
Status: Completed | Type: Observational
Sponsor: University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, Dr. Wolfgang Bömicke, Principal Investigator, University Hospital Heidelberg
Other Study IDs: ZI²
Record Dates: First submitted 2021-08-10; First posted 2021-09-02 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Jaw, Edentulous; Dental Impression Techniques
Keywords: intraoral scan; scanning accuracy; edentulousness; implant scan; digital impression
MeSH Terms: conditions — Jaw, Edentulous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Locator Group: The participant has a mandibular overdenture supported by two implants with locator attachments. The implants are scanned with each of two intraoral scanners both with and without the use of artificial landmarks. The implant scans are analyzed in terms of scanning accuracy (trueness and precision) by comparison with a reference model (3D implant positions in the working cast of the immediately loaded overdenture).
- Bar Group: The participant has a mandibular overdenture supported by two implants with a dolder bar attachment. The implants are scanned with each of two intraoral scanners both with and without the use of artificial landmarks. The implant scans are analyzed in terms of scanning accuracy (trueness and precision) by comparison with a reference model (3D implant positions in the working cast of the immediately loaded overdenture).

SUMMARY:
Today, tooth- or implant-supported single crowns and short-span fixed partial dentures can be fabricated on the basis of an intraoral scan, but the scanning accuracy decreases with increasing length of the jaw section to be captured. An accurate scan is also made more difficult by edentulous jaw sections, as these provide the scanner with few landmarks for proper three-dimensional image composition.

With respect to both edentulous and edentulous patients with dental implants, the currently available literature does not provide a firm basis for deciding whether such patients can already be scanned with sufficient accuracy. It is considered problematic in this context that the findings on digital impression accuracy, regardless of whether teeth or implants have been scanned, are based almost exclusively on the results of in vitro studies. Conclusions about the accuracy of intraoral scanners under clinical conditions with moving patients and limited accessibility to the structures to be imaged, especially in the presence of blood, saliva or sulcus fluid, are extremely limited based on these data.

Therefore, the aim of this study is to determine the clinical scanning accuracy of two current intraoral scanning systems for the three-dimensional acquisition of the position of two interforaminal dental implants in the edentulous mandible. The influence of artificial landmarks to achieve increased scan accuracy will also be tested.

ELIGIBILITY:
Inclusion Criteria:

* Participants who had received a mandibular overdenture supported by two implants with either Locator attachments or a Dodler bar attachment following an immediate loading protocol as part of a randomized controlled trial [Kappel S, Giannakopoulos NN, Eberhard L, Rammelsberg P, Eiffler C. Immediate Loading of Dental Implants in Edentulous Mandibles by Use of Locator® Attachments or Dolder® Bars: Two-Year Results from a Prospective Randomized Clinical Study. Clin Implant Dent Relat Res. 2016 Aug;18(4):752-61. doi: 10.1111/cid.12349. Epub 2015 May 7. PMID: 25950679.] and for whom intact working casts with laboratory implant analogs representing the reference implant positions were available.
* Participant is legally capable
* Signed informed consent form available

Exclusion Criteria:

* Participant not contactable
* Participant not willing to participate
* New overdenture or dolder bar attachment based on a working cast other than that used for immediate loading
* No intact working casts available
* Diagnosed epilepsy
* Pregnancy and lactation
* Local or systemic acute or chronic (also in the past) general medical diseases and conditions, which contradict a participation in the study and or expose the patient to a higher risk in case of a study participation
* Known allergies or intolerances to the materials used in the study.
* Lack of compliance

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants had received a mandibular overdenture supported by two implants with either Locator attachments or a Dodler bar attachment following an immediate loading protocol as part of a randomized controlled trial [Kappel S, Giannakopoulos NN, Eberhard L, Rammelsberg P, Eiffler C. Immediate Loading of Dental Implants in Edentulous Mandibles by Use of Locator® Attachments or Dolder® Bars: Two-Year Results from a Prospective Randomized Clinical Study. Clin Implant Dent Relat Res. 2016 Aug;18(4):752-61. doi: 10.1111/cid.12349. Epub 2015 May 7. PMID: 25950679.].
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Effect of intraoral scanner on scanning accuracy | through study completion, an average of 2 hours
  Accuracy will be given as trueness and precision according to ISO 20896-1:2019 Dentistry - Digital impression devices - Part 1: Methods for assessing accuracy. Implant distance deviations will be measured in [µm] and implant angle deviations in [°].

SECONDARY OUTCOMES:
Effect of artificial landmarks on scanning accuracy | through study completion, an average of 2 hours
  Accuracy will be given as trueness and precision according to ISO 20896-1:2019 Dentistry - Digital impression devices - Part 1: Methods for assessing accuracy. Implant distance deviations will be measured in [µm] and implant angle deviations in [°].
Effect of implant attachment on scanning accuracy in [µm] and [°] | through study completion, an average of 2 hours
  Accuracy will be given as trueness and precision according to ISO 20896-1:2019 Dentistry - Digital impression devices - Part 1: Methods for assessing accuracy. Implant distance deviations will be measured in [µm] and implant angle deviations in [°].
Effect of intraoral scanner/use of artificial landmarks on intraoral scanning process/quality of the 3D dataset by a study investigator on the basis of qualitative criteria (see description) | through study completion, an average of 2 hours
  Effect of intraoral scanner/use of artificial landmarks on intraoral scanning process (successful, successful with difficulties, failed)/quality of the 3D dataset (Surface irregularities, deformations, stitching errors, other)

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Bömicke, Prof. Dr., Principal Investigator — Department of Prosthetic Dentistry, University of Heidelberg
Locations (1):
- Department of Prosthetic Dentistry, University Hospital Heidelberg, University of Heidelberg, Heidelberg, Baden-Wurttemberg, Germany